CLINICAL TRIAL: NCT04878016
Title: A Phase III, Randomized，Double-blind Placebo-controlled Study of Carboplatin Plus Etoposide With or Without ZKAB001 (Anti-PD-L1 Antibody) in Patients With Untreated Extensive-stage Small Cell Lung Cancer
Brief Title: A Study of Carboplatin Plus Etoposide With or Without ZKAB001 (Anti-PD-L1 Antibody) in Patients With ES-SCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZKAB001-LEES-2020-07
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZKAB001＋carboplatin+etoposide (Experimental): The induction phase will consist of four cycles of ZKAB001 plus chemotherapy, with each cycle being 21 days in duration. On Day 1 of each cycle, patients will receive drug infusions in the following order:
  ZKAB001 → carboplatin → etoposide
  Interventions: Biological: ZKAB001; Drug: Carboplatin; Drug: Etoposide
- placebo + carboplatin + etoposide (Placebo Comparator): The induction phase will consist of four cycles of placebo plus chemotherapy, with each cycle being 21 days in duration. On Day 1 of each cycle, all eligible patients will receive drug infusions in the following order:
  placebo → carboplatin → etoposide
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Biological: ZKAB001 — Patients will receive ZKAB001 5mg/kg administered by IV infusion every 21days，
  Arms: ZKAB001＋carboplatin+etoposide
Drug: Placebo — Patients will receive placebo administered by IV infusion every 21days.
  Arms: placebo + carboplatin + etoposide
Drug: Carboplatin — Carboplatin should be administered after completion of placebo/ZKAB001 by IV infusion over 30-60 minutes to achieve an initial target AUC of 5 mg/mL/min. Carboplatin and etoposide will be used for a total of 4 cycles， followed by placebo/ZKAB001 maintenance therapy.
Drug: Etoposide — Etoposide (100 mg/m^2) should be administered intravenously over 60 minutes following carboplatin administration. On Days 2 and 3 of each cycle, etoposide 100 mg/m2) should be administered intravenously over 60 minutes.
  Carboplatin and etoposide will be used for a total of 4 cycles， followed by placebo/ZKAB001 maintenance therapy.

SUMMARY:
This is a randomized, Phase III, multicenter, double-blinded, placebo-controlled study designed to evaluate the safety and efficacy of ZKAB001 in combination with carboplatin + etoposide compared with treatment with placebo + carboplatin + etoposide in patients who have ES-SCLC and are untreated for their extensive-stage disease.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled multicenter III study.

Eligible patients will randomly enter the trial group or control group at 1:1, that is, ZKAB001+ carboplatin + etoposide or placebo + carboplatin + etoposide, with a treatment cycle every 3 weeks. There are 4 cycles of chemotherapy.

Stratification factors included gender (male / female), PS score (0/1) and brain metastasis (yes / no).

The study included screening period, treatment period (subjects received study treatment until confirmed disease progression, or intolerable toxic reaction, or reached the maximum medication cycle of 2 years, or the subject voluntarily requested the end of the study treatment) and follow-up period (including safety follow-up and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women, age ≥ 18 years.
2. Small Cell Lung Cancer confirmed by histology or cytology.
3. Extensive-stage SCLC (defined as AJCC 8th Edition IV (Tany,Nany,M1a/b/c), or T3-4 cannot be included in a tolerable radiotherapy plan due to multiple pulmonary nodules or tumor/nodule size).
4. Have not received first-line systemic treatment for ES-SCLC in the past.
5. surgery and adjuvant therapy for cure, such as radiotherapy and chemotherapy, were performed in the past, and there was no treatment interval of at least 6 months from the last chemotherapy, radiotherapy or radiotherapy or chemotherapy to the diagnosis of ES-SCLC.
6. ECOG PS 0,1.
7. The estimated survival ≥ 8 weeks.
8. CT or MRI scan with at least one measurable lesion (according to RECIST v1.1) ≤ 28 days before administration of the first study drug.
9. Male partners of childbearing age and female subjects of childbearing age must have contraception within 6 months after signing the informed consent form to the last study of the drug, and the (HCG) test of human chorionic gonadotropin in blood / urine of female subjects of childbearing age must be negative 7 days before the first use of the drug.
10. Before the first dose , the laboratory test values meets the following conditions: (1) Blood routine test (corrected without blood transfusion and hematopoietic factor drugs within 14 days before screening): White blood cell count ((WBC) ≥ 3.0x10^9); absolute neutrophil count ((ANC)) ≥ 1.5x10^9; platelet (PLT) ≥ 100x10^9; hemoglobin content ((hGB) ≥ 90g). (2) Liver function: aspartate aminotransferase (AST) ≤ 2.5 ULN, alanine liver aminotransferase (ALT) ≤ 2.5 ULN; ALT and AST < 5 ULN; serum total bilirubin (TBIL) ≤ 1.5 ULN; albumin (ALB) ≥ 30 g L; (3) Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance rate (Ccr) ≥ 40 mL/min (Cockcroft/Gault formula). (4) Coagulation function: international standardized ratio (INR) ≤ 1.5 ULN, activated partial thromboplastin time (APTT) ≤ 1.5 ULN; (5) alkaline phosphatase (ALP) ≤ 2.5 ULN, bone metastasis subjects, ALP ≤ 5 ULN.
11. Tumor tissue samples that can meet the the requirements of PD-L1 expression detection can be provided within 4 weeks from the screening period to 4 weeks after enrollment.
12. Sign informed consent form voluntarily，have good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Received any T cell costimulatory or immune checkpoint inhibitors before entering the group, including, but not limited to, cytotoxic T lymphocyte associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other drugs targeting T cells; previously received anti-vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR) therapy.
2. Active brain metastasis or meningeal metastasis. Patients with brain metastasis after treatment need to meet the following conditions: asymptomatic; no imaging evidence of progress ≥ 4 weeks after treatment; completion of treatment within 7 days before the first dose of the study drug; and no need to receive systemic corticosteroids (> 10mg/ prednisone or equivalent) less than 14 days before the first dose of the study drug. If a new asymptomatic brain metastasis is found during the screening period, radiotherapy and/or surgery are required.

   If all other criteria are met after treatment, additional brain scans are not required before randomization.
3. The completion time of radiotherapy for the brain and palliative radiotherapy for the focus of bone disease is less than 7 days before the first dose of the study drug.
4. Active, known or suspected autoimmune diseases, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granuloma, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis. Only cases of residual hypothyroidism due to autoimmune thyroiditis, controlled type I diabetes, or no recurrence expected in the absence of external stimulation that require hormone replacement therapy can be included. Only patients with eczema, psoriasis, neurodermatitis or vitiligo (psoriatic arthritis patients will need to be excluded) can be enrolled in the group if they meet the following conditions: the area covered by the rash must be less than 10% of the body surface area; the disease is well controlled at the baseline level, requiring only inefficient topical steroids, and those with no acute exacerbation in the past 12 months can be enrolled.
5. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage (once a month or more frequently). Patients who use indwelling catheters are allowed to be selected.
6. Corticosteroids (> 10 mg/ prednisone or equivalent dose) or other immunosuppressants were used within 14 days before the first study. Inhalation or topical use of steroids and adrenal replacement steroids are allowed in the absence of active autoimmune disease; for patients receiving short-term, systemic immunosuppressive therapy, for example, glucocorticoids for nausea, vomiting, or allergic reaction management or preventive use can be admitted after consultation with the sponsor. Allow the use of salt corticosteroids in the treatment of postural hypotension and the use of low-dose glucocorticoid supplements in the treatment of adrenocortical insufficiency.
7. Patients who had been vaccinated or planned to receive live vaccines within 4 weeks before drug administration were studied for the first time.
8. Major surgery was performed within 4 weeks before drug administration, or major surgery was planned during the study period.
9. Interstitial pneumonia (ILD) disease, drug-induced pneumonia, radiation pneumonia requiring steroid treatment or active pneumonia with clinical symptoms.
10. Active pulmonary tuberculosis or screening patients with a history of active pulmonary tuberculosis infection within 1 year before treatment, whether treated or not.
11. Uncontrolled cardiovascular diseases, such as: (1) New York Heart Association (NYHA) grade 2 or above heart failure (2) unstable angina pectoris (3) myocardial infarction or cerebrovascular accident within 6 months (4) clinically significant supraventricular or ventricular arrhythmias need to be treated.
12. Uncontrolled active infections (e.g. need intravenous antibiotics, antifungal or antiviral therapy).
13. Active hepatitis B or C (unless HBV-DNA titer < 500IU/mL or copy number < 1000copies/ml, HCV-RNA negative after antiviral treatment can be included in), HIV positive or known history of acquired immunodeficiency syndrome.
14. Known allergies to research drugs or excipients, and known severe allergic reactions to any monoclonal antibody; allergic history of carboplatin or etoposide.
15. Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation.
16. Other malignant tumors occurred less than 5 years before the first dose, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical mastectomy.
17. Have been treated with any other experimental drugs or participated in another interventional clinical study within 4 weeks before signing ICF.
18. Pregnant or lactating women.
19. Known cases of mental illness, alcohol abuse, inability to quit smoking, drug use or substance abuse.
20. Other situations judged by the investigators to be unsuitable for inclusion in the group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years
  The time from the date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
progression free survival | 2 years
  The time between the date of randomization and the date of first documented disease progression or death, whichever occurs first.
objective response rate | 2 years
  ORR is defined as either an unconfirmed CR or a PR, as determined by the investigator using RECIST v1.1.
disease control rate | 2 years
  It refers to the percentage of patients with the best overall efficacy of CR, PR and SD and maintained for more than 4 weeks in patients who can evaluate the efficacy.
duration of response | 2 years
  DOR is defined as the time interval from the date of the first occurrence of a CR or PR (whichever status is recorded first) until the first date that progressive disease or death is documented, whichever occurs first.
Time to Deterioration | 2 years
  Time to deterioration will be measured using the EORTC QLQ-C30.
Time to Deterioration | 2 years
  Time to deterioration will be measured using the EORTC QLQ-LC13.
Safety Outcome Measures | 2 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Z, Chen J, Huang D, Zhang W, Wu L, Yi T, Wang Q, Han L, Tan L, Li Y, Zhang Z, Li N, Li J, Zhang T, Hu Y, Sun H, Wu Y, He Z, Yang R, Cheng P, Li X, Shi J, Yu G, Ma D, Li BX, Dai X, Wong M, Li Y, Yu X, Lu S; Socazolimab Study Group. A multicenter, randomized, double-blind, placebo-controlled phase 3 study of Socazolimab or placebo combined with carboplatin and etoposide in the first-line treatment of extensive-stage small cell lung cancer. Signal Transduct Target Ther. 2025 Jan 13;10(1):28. doi: 10.1038/s41392-024-02115-5. PMID 39800716
- [Derived] Lu S, Chen Z, Cui J, Guo R, Li Z, Li BX, Dai X. Efficacy and Safety of Anti-Programmed Death-Ligand 1 Monoclonal Antibody Socazolimab With Carboplatin and Etoposide for Extensive-Stage SCLC: Results From the Phase 1b Clinical Trial. JTO Clin Res Rep. 2023 Feb 28;4(4):100478. doi: 10.1016/j.jtocrr.2023.100478. eCollection 2023 Apr. PMID 37020926